CLINICAL TRIAL: NCT06971913
Title: Efficacy and Safety of Low-dose IL-2 in SLE Patients With CMV Viremia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, He Jing, PhD, MD, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLE-CMV-IL2
Record Dates: First submitted 2025-02-18; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: SLE (Systemic Lupus); CMV
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Interleukin-2; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IL-2 group (Experimental): IL-2 group are going to be treated with low-dose IL-2 plus ganciclovir.
  Interventions: Drug: Interleukin-2 (IL-2); Drug: Ganciclovir (GCV)
- Control group (Other): Control group will be treated with ganciclovir until negative test for CMV DNA load
  Interventions: Drug: Ganciclovir (GCV)

INTERVENTIONS:
Drug: Interleukin-2 (IL-2) — Low-dose IL-2 at 1MIU will be administered subcutaneously every other day from baseline to CMV negativity.
  Arms: IL-2 group
Drug: Ganciclovir (GCV) — Ganciclovir injection will be administrated intravenously at a dose of 5mg/kg per day.

SUMMARY:
This clinical trial will assess the efficacy and safety of low-dose interleukin-2 (IL-2) treatment in systemic lupus erythematosus (SLE) complicated with cytomegalovirus (CMV) viremia.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune syndrome affecting various organs, and infection is the leading cause of death in SLE. SLE patients are prone to opportunistic infections such as CMV viremia due to treatments with glucocorticoids and immunosuppressives. CMV viremia is a life-threatening complication in the immunocompromised population, which could establish a state of long-term latency following infection. Once CMV is reactivated in hosts, the immune system would be attacked, resulting in exacerbating SLE disease condition.

While traditional available therapies for SLE patients with CMV viremia, to a certain extent, have improved the outcome of these patients, there remains many patients who are antiviral drug-resistant or nonresponsive in clinical practice. Thus, there is an unmet need for safe and more effective treatments. In preliminary clinical trials, we have demonstrated low-dose IL-2 is safe and efficient in autoimmune diseases, including rheumatoid arthritis and SLE. In addition, in spite of sacrificing anti-infection immune function as most immunosuppressive drugs, low-dose IL-2 therapy lowered incidence of infections by upregulating the level of natural killer (NK) cells in SLE patients. In addition, low-dose IL-2 therapy is much less economically burdensome than intravenous immunoglobulin. We hypothesized that low-dose IL-2 could be a novel therapy in SLE patients with CMV viremia.

This is a multicenter, prospective and controlled study to evaluate the efficacy/safety of low-dose IL-2 plus ganciclovir in SLE with active CMV infection.

Methods: SLE patients with CMV viremia will be enrolled and randomly assigned (1:1 ratio) to two groups, low-dose IL-2 group or control group in this study. IL-2 group are going to be treated with low-dose IL-2 plus ganciclovir. Low-dose IL-2 at 1MIU will be administered subcutaneously every other day from baseline to CMV negativity. Ganciclovir injection will be administrated intravenously at a dose of 5mg/kg per day. Control group are going to be treated with ganciclovir. Weekly follow-ups visits will be conducted until participants became CMV negative, the criteria for withdrawing from the trial. The endpoints were changes in NK cells, duration of CMV viremia, clinical, immunologic responses and safety.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology criteria for the diagnosis of SLE.
* The test for plasma CMV DNA viral load is positive.
* Age: 18 to 65 years, weight 45-80kg, male or female, gender ratio is not limited.
* Apply corticosteroid less than 1.0mg/kg/d.
* Written informed consent form.

Exclusion Criteria:

* Inability to comply with IL-2 treatment regimen;
* Other active infections. (hepatitis B or C virus, Epstein-Barr virus, human immunodeficiency virus, Mycobacterium tuberculosis or pneumocystis carinii pneumonia)
* Any anti-CMV vaccine within 6 months;
* History of intravenous immunoglobulin (IVIG) or leflunomide within 6 months prior to randomization, and those who have undergone plasmapheresis;
* Active severe neuropsychiatric manifestations of SLE;
* Severe chronic liver, kidney, lung or heart dysfunction; (heart failure (≥ grade III NYHA), hepatic insufficiency (transaminases> 3N));
* Severe complications. (respiratory failure, heart failure or toxic shock)
* Complicated with other autoimmune diseases;
* Cancer or history of cancer cured for less than five years (except in situ carcinoma of the cervix or Basocellular carcinoma);
* Pregnancy or lactation in females.
* Mental disorder or any other chronic illness or drug-abuse that could interfere with the ability to comply with the protocol or to give information;
* Participate in other clinical trial within 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes of NK cell levels | Baseline and week 12
  Changes of absolute NK cell count and NK%.

SECONDARY OUTCOMES:
Duration of CMV viremia | From enrollment to the end of treatment
  Duration of CMV viremia is defined as the time interval between detection of positive CMV DNA load in plasma and CMV negativity.
Change of CMV titers | From enrollment to the end of treatment
  The change (decline) of CMV titers from baseline
Immune responses | Baseline and Week 12
  Changes of levels of immunoglobulins and lymphocyte subtypes, including T/B lymphocytes, Treg, Th1/2/17.
• Complements levels | Baseline and week 12
  Changes of levels of complement 3/4 (C3/C4)
Adverse events (AEs) | Baseline and week 12
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Bejing, China